CLINICAL TRIAL: NCT06283381
Title: Effect of Proton Pump Inhibitors on the Structural Integrity of Endoscopic Sleeve Gastroplasty: a Single-centre Open-label, Randomized, Controlled Pilot Clinical Trial
Brief Title: The ESG Integrity Study: Effect of Proton Pump Inhibitors on the Structural Integrity of Endoscopic Sleeve Gastroplasty
Acronym: ESGIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4264
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: experimental group (Experimental): no administration of Esomeprazole or any other proton pump inhibitor after the Endoscopic Sleeve Gastroplasty
  Interventions: Drug: Esomeprazole
- Arm B: standard of care group (Active Comparator): administration of Esomeprazole 40 mg twice a day for 4 weeks and 40 mg once a day for another 4 weeks after the Endoscopic Sleeve Gastroplasty
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — oral administration, tablets, 40 mg

SUMMARY:
The study is a single center randomized, open-label, phase IV clinical trial. Obese patients who have indication to Endoscopic sleeve gastroplasty (ESG) for clinical reasons are included and ESG is performed as per clinical practice. After randomization, the patients are divided in two arms:

* Arm A: patients will stop proton pump inhibitors (PPI) 24h after the procedure.
* Arm B: patients will assume oral Esomeprazole 40 mg twice a day for 4 weeks and 40 mg once a day for 4 weeks (total 8 weeks of PPIs after ESG- standard current treatment).

The primary aim of the study is to evaluate the effect of PPI on the structural integrity of the ESG

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 65 years
* BMI between 30 to 45 kg/m2
* Willingness to participate in the study and ability to comply and understand the study protocol.

Exclusion Criteria:

* Active gastric gastro-duodenal during the last 6 months
* Helicobacter pylori infection.
* Organic or motility disorder of the stomach and / or esophagus
* Anticoagulant treatment
* Previous bariatric surgery or any other type of surgery of the esophagus, stomach and duodenum
* Ongoing or active malignancy during the last 5 years.
* Myocardial infarction during the past 6 months or/and heart failure class III or IV according to the New York Heart association's classification.
* Drug or alcohol abuse
* Bulimic or binge eating pattern
* Continuous glucocorticoid or anti-inflammatory treatment
* Uncontrolled thyroid disease.
* Pregnancy, breastfeeding
* Psychiatric or cooperative problems or low compliance that is a contraindication from participating in the study.
* Hiatal hernia ≥ 5 cm
* Known allergy or hypersensitivity to the active substance or any of the other excipients
* Liver cirrhosis of any Child-Phugh stage or MELD> 15
* Chronic Severe Renal Insufficiency (eGFR < 30 ml/min/1.73 m2 based on CKD-EPI equation)
* Currently participating in other study, or previously participated in an experimental drugs trial within 30 days before or 5 half-life of the drug administered
* Any health issue that might put the patient at risk if the treatment is performed, judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The structural integrity of the sutures after Endoscopic sleeve gastroplasty (ESG) | 6 months
  The structural integrity of the ESG will be defined as opened (all stitches loose), partially intact (at least one stitch loose), or intact (all stitches tight).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy